CLINICAL TRIAL: NCT05515367
Title: A Phase 4,52 Week, Single Arm,Multicentre Post Marketing Surveillance to Evaluate the Safety of Desidustat for the Treatment of Anemia in Subjects With Chronic Kidney Disease (CKD).
Brief Title: A Post Marketing Surveillance to Evaluate the Safety of Desidustat for the Treatment of Anemia in Subjects With Chronic Kidney Disease (CKD).(Real World Evidence Study)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DESI.22.001
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Diseases; Anemia of Chronic Kidney Disease
Keywords: Real World Evidence Study
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — desidustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Desidustat oral tablet (Experimental): Oral administration of Desidustat from baseline (week 0) to Week 52
  Interventions: Drug: Desidustat

INTERVENTIONS:
Drug: Desidustat — Oral tablet

SUMMARY:
A Phase 4, 52 week, single arm, multicentre post marketing surveillance to evaluate the safety of Desidustat for the treatment of anemia in subjects with chronic kidney disease (CKD)

DETAILED DESCRIPTION:
The study is being planned to evaluate long term safety of Desidustat with CKD patient.

Total 1004 population i.e 502 dialysis dependent, 502 dialysis independent.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age.
2. Current clinical diagnosis of anemia due to CKD, baseline hemoglobin concentrations must be 7.0-11.0 g/dL (both inclusive) before the enrolment.
3. Ability to understand and give informed consent for participation.
4. No significant folate or Vitamin B12 deficiency.
5. Females of childbearing potential, must agree to use one of the approved contraception methods, from screening until End-of-study visit.
6. For Subjects dependent on hemodialysis:

   1. Must be receiving haemodialysis session ≥2 times in a week for at least 12 weeks prior to screening visit and have access consisting of an arteriovenous fistula, AV graft, or catheter (permanent/temporary).
   2. Subjects will be considered not treated with erythropoietin analogue (Epoetin and Darbepoetin) if they have not received erythropoietin analogue for at least 4 weeks and Mircera® for at least 8 weeks prior to screening visit. OR Subjects who are on ESA therapy must be on stable dose for 4 weeks prior to enrolment (≤30% of dose change).

Exclusion Criteria:

1. Subjects who received red blood cell transfusion within 8 weeks prior to enrolment.
2. Pre-dialysis subjects, who had prior exposure to ESA agents within 6 weeks prior to enrolment.
3. In case of diabetes mellitus subjects, glycosylated haemoglobin (HbA1c) > 9 %.
4. In case of hypertensive subjects, systolic and diastolic BP (Blood pressure) is >160 and 100 mm of Hg respectively or uncontrolled blood pressure.
5. History of previous or concurrent cancer or renal transplant or severe allergic or hypersensitivity to investigational products and its excipients or chronic inflammatory disease (RA, Celiac disease, UC, Crohn's disease, Systemic Lupus Erythematosus [SLE]).
6. Serologic status reflecting active Hepatits B or C infection or Human Immunodeficiency virus (HIV) infection.
7. History of uncontrolled autoimmune haemolytic anemia, idiopathic thrombocytopenic purpura (ITP) or thalassemia/bleeding disorders or clinical conditions (e.g. gastrointestinal [GI] bleeding or constitutional disorders) that may increase risk of life-threatening bleeding./ requires or is receiving anticoagulation with warfarin or equivalent vitamin K antagonists or other medications within 28 days of the first dose of study drug that in the investigator's opinion, could compromise subject safety.
8. Major surgery within 90 days and minor surgery within 30 days prior to the enrolment of the subject.
9. Unable to swallow tablets or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption such as; mal-absorption syndrome, resection of the small bowel or poorly controlled inflammatory bowel disease affecting the small intestine.
10. History of myocardial infarction or stroke or intracranial haemorrhage within 6 months prior to enrolment.
11. Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, any class 3 or 4 cardiac disease as defined by the NYHA (New York Heart Association) classification.
12. Current life-threatening illness, medical condition, systemic disorders (e.g., respiratory, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or any other body system involvement) or laboratory abnormalities which, in the Investigator's opinion, could compromise the subject's safety.
13. History of significant alcoholism or drug abuse within the past 1 year. History or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco/nicotine products (more than 10 times per day).
14. History of difficulty with donating blood.
15. History or presence of any clinically significant ECG abnormalities during screening.
16. Participants who have participated in any drug research study other than the present trial within past 3 months.
17. Female volunteers with following criteria will not be eligible:

    1. History of pregnancy or lactation in the past 3 months.
    2. Fertile female volunteers not protected against pregnancy by adequate long-term anti-fertility measures.
    3. History of less than 1 year of menopause and not using adequate long-term antifertility measures.
    4. Oral hormone replacement therapy.
    5. Positive serum β-hCG level at the screening visit.
    6. Pregnant and breastfeeding women.
18. Abnormal baseline laboratory investigations as follows:

    1. WBC count ≤3 x 103/μL.
    2. Platelets count ≤100 x 103/μL.
    3. Bilirubin ≥2.0 mg/dL.
    4. ALT and/or AST ≥2.5 times of the ULN.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
To asses the Proportion of Subjects with treatment emergent adverse events. | Baseline (week 0) to Week 52 (end of treatment)
To asses the Proportion of Subjects with treatment emergent Serious adverse events. | Baseline (week 0) to Week 52 (end of treatment)

SECONDARY OUTCOMES:
Mean change in hemoglobin level | Baseline (week 0) to Week 52 (end of treatment)
Mean change in Lipid profile including Small dense LDL from baseline | Baseline (week 0) to Week 52 (end of treatment)
Mean change in VEGF | Baseline (week 0) to Week 52 (end of treatment)
Mean change in serum Hepcidin | Baseline (week 0) to Week 52 (end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Deven Parmar, MD,FCP, Study Chair — Zydus Therapeutics Inc.
Locations (1):
- Indira Gandhi Institute of Medical Sciences, Sheikhpura, Bihar, India

IPD SHARING:
Plan to Share IPD: No